CLINICAL TRIAL: NCT07406061
Title: Multi-Dimensional, Real-time Ultrasound Imaging of the Head, Neck, and Airway
Brief Title: Ultrasound Imaging of the Head, Neck, and Airway
Status: Not yet recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00116760
Record Dates: First submitted 2026-01-09; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: Ultrasound; Upper airway; ultrasonography
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Simple ultrasonography imaging

SUMMARY:
Purpose and Objectives: The main purpose is to test an ultrasound device that can assess the upper airway to create dynamic 4D imaging, which current technology cannot do. Ultrasound waves travel well within soft tissue but are unable to penetrate cartilage, bone, and air-filled structures, obscuring findings which are covered by these structures and limiting the ability of the ultrasound to adequately image posterior to the soft tissue upper airway, trachea, or behind the mandible.

DETAILED DESCRIPTION:
Ultrasound has been used clinically for over 50 years and it is now the most common imaging method for cardiac and abdominal imaging in the world. Ultrasound system development using phased array techniques began at Duke almost 45 years ago with Duke system, referred to as T1: the T standing for Thaumascan, an early name for the Duke system. Virtually all current ultrasound scanners in the world today use the same basic phased array technology pioneered at Duke using the T1 (and its progeny) device(s). This family of ultrasound systems has been developed in the Department of Biomedical Engineering in collaboration with the Division of Cardiology.

T5 is a high-speed, real-time, 32:1 parallel processed, 2D and 3D ultrasound imaging scanner connected to a 4000 element matrix array, of which 1280 elements are actively used (up to 512 independent transmitters and 1024 independent receivers). The system is capable of acquiring high-speed B- and C-mode grey scale images, real-time orthogonal and parallel images and real-time 2D and 3D ultrasound images. The system is unique in that its components are highly configurable to allow for a variety of different parameter settings to derive the best image quality possible. Uniquely, T5 can image synchronously with multiple transducers at spatially different locations.

This protocol is intended to provide for system modification and initial testing of new ultrasound methods. Changes in the system will be determined mainly by the subjective results of initial or periodic scanning. The first step in this process requires establishing whether head, neck, and airway images are even possible in certain scanning configurations. Included in this is learning how to scan with the device. The second step will determine various subjective image quality comparisons (one system configuration against another). Image quality is determined by assessing system capability for target acquisition, gray scale, and resolution in the resulting images. The third step can be undertaken when adequate images are available. Here, subjective comparisons of results from T5 will be made against those from other conventional imaging methods otherwise obtained in the regular course of a subject's care (as they are available).

This project is investigator funded. It is hoped that the results of this study will be instrumental in the initiation of the applications for funding from governmental or other agencies.

There is broad agreement that ultrasound involves only minimal subject risk. Diagnostic ultrasound imaging from the body surface has been cited by the FDA as an example of a non-significant risk study in the "Investigational Device Exemptions Manual" June, 1996, HHS Publication FDA 96-4159. The transducer in the Duke system uses conventional levels of ultrasound energy, and is at, or below, the ultrasound energy in use today in commercial systems and approved by the Food and Drug Administration (720 mW/cm ; M. 2 I. = 1.9). Thus, there is no added patient risk in the use of this device when compared to conventional ultrasound scanning. Whatever the scanning configurations, the power output of the machine does not increase.

This protocol provides for the acquisition of images of the upper airway to initially establish, then progressively improve, Duke T5 ultrasound system performance in a stepwise fashion. Understanding the purpose and execution of this protocol requires the understanding of the stepwise and iterative processes of:

Step 1: development of scanning procedures Step 2: image improvement Step 3: exploration of image comparisons in small groups of patient

ELIGIBILITY:
Inclusion Criteria:

* Capable of lying stationary in a supine position for the duration of the stud

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers ages 18 or higher
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Tracheal diameter (mm) | Day 1
  Ultrasound will be used to scan the exterior of the neck and submandibular region to assess airway dimensions in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Initially the data will be reviewed and analyzed before considering sharing.